CLINICAL TRIAL: NCT01394237
Title: Laparoscopic Sacrocolpopexy: Long Term Results With Special Focus on Anatomical Results and Quality of Life
Brief Title: Laparoscopic Sacrocolpopexy: Long Term Follow-up
Status: Completed | Type: Observational
Sponsor: Kantonsspital Aarau (Other)
Responsible Party: Principal Investigator, Dimitri Sarlos, Head Gynaecology and oncological Gynaecology, Kantonsspital Aarau
Other Study IDs: SakPexFup
Record Dates: First submitted 2011-07-13; First posted 2011-07-14 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-03

CONDITIONS: Vaginal Vault Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Operated by laparoscopic sacrocolpopexy: Patients operated at our institution by laparoscopic sacrocolpopexy between 2003 and 2007
  Interventions: Other: Examination

INTERVENTIONS:
Other: Examination — Examination of recurrences of vaginal vault prolapse measured as objective anatomical results using the pelvic organ prolapse quantification (POP-Q) system
  Other Names: exam; test; assessment

SUMMARY:
The purpose of this study is to determine the long term results of laparoscopic sacrocolpopexy regarding anatomical results, recurrences, complications, further surgeries required, patients satisfaction and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated for vaginal vault prolapse at our institution by laparoscopic sacrocolpopexy between 2003 and 2007
* consent

Exclusion Criteria:

* no consent

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated for vaginal vault prolapse at our institution by laparoscopic sacrocolpopexy between 2003 and 2007
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Recurrences according to pelvic organ prolapse quantification (POP-Q) assessment | 3-6 years after surgery
  Recurrences of vaginal vault prolapse measured as objective anatomical results using the pelvic organ prolapse quantification (POP-Q) system

SECONDARY OUTCOMES:
Quality of life | 3-6 years after surgery
  Quality of life as assessed by a specific validated questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Sarlos, MD, Study Director — Kantonsspital Aarau
Locations (1):
- Frauenklinik Kantonsspital Aarau, Aarau, Canton of Aargau, Switzerland

REFERENCES:
- [Background] Sarlos D, Brandner S, Kots L, Gygax N, Schaer G. Laparoscopic sacrocolpopexy for uterine and post-hysterectomy prolapse: anatomical results, quality of life and perioperative outcome-a prospective study with 101 cases. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Oct;19(10):1415-22. doi: 10.1007/s00192-008-0657-0. Epub 2008 Jun 7. PMID 18536861